CLINICAL TRIAL: NCT02674997
Title: A New Patient-centric Outcome Measure for Patients With Hemophilia: Testing the Feasibility of GAS-Hem in Pediatric, Adolescent and Adult Hemophilia A Patients
Brief Title: GAS-Hem Feasibility Study
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 001501
Record Dates: First submitted 2015-11-24; First posted 2016-02-05 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia A
Keywords: Goal setting; Feasibility; Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem); Patient reported outcome (PRO); Goal attainment scaling (GAS)
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study participants: Participants with Hemophila A
  Interventions: Biological: Factor VIII

INTERVENTIONS:
Biological: Factor VIII — Licensed Factor VIII products. Study is brand agnostic
  Other Names: FVIII

SUMMARY:
The purpose of this study is to investigate the feasibility and acceptability of the Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) as a patient reported outcome (PRO) measure to monitor clinical progress in participant-identified goal areas in individuals with hemophilia A.

DETAILED DESCRIPTION:
Hemophilia A is an X-linked recessive, congenital bleeding disorder caused by deficient or defective coagulation factor VIII (FVIII). The absence of FVIII leads to 'spontaneous' bleeding episodes (occurring primarily in joints, muscles and, less commonly, in soft tissues) and to excessive bleeding following trauma or injury. With proper treatment (FVIII) and self-care, most hemophilia patients can maintain an active, productive lifestyle. With a growing appreciation that a low bleed rate sometimes is only achieved, in part, by patients limiting their activities, there has been growing interest in understanding how hemophilia may still limit life despite absence of major bleeds. The current study will introduce and test a standardized method for individualized outcome measurement based on Goal Attainment Scaling (GAS), a method that allows participants to set goals to address challenges that are meaningful to them and monitor attainment in those areas over time. The Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) is an online instrument for setting and tracking personalized goals related to hemophilia. The goal menu captures common challenges faced by people with hemophilia, accompanied by an inventory of descriptors that can be personalized. The tool can be used to track the health of individuals across a wide spectrum of ages, life experiences and health states. This is a 12-week, multicenter, prospective, observational, feasibility study of up to 60 people (aged 5 and 65) with moderate to severe hemophilia A to investigate the feasibility and acceptability of GAS-Hem as a patient reported outcome (PRO) measure to monitor clinical progress in participant-identified goal areas. Outcomes, including GAS-Hem (primary), health-related quality of life, bleeding episodes (location, cause, time) and treatment (time, dose and reason for infusion) will be assessed at screen/baseline, with follow-up at 6 and 12 weeks. Endpoints of interest include participant GAS-Hem outcomes at 6 and 12 weeks, participant quality of life (QoL) outcomes at 6 and 12 weeks, as well as participant and clinician perception of the GAS-Hem as a useful means of identifying and monitoring progress in relevant goal areas.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a documented diagnosis of hemophilia A
2. Participant has documented clotting factor levels of 5% or less
3. Participant is on a prescribed regimen of continuous prophylaxis. Continuous prophylaxis is defined by the World Federation of Hemophilia as "… the intent of treating for 52 weeks a year and receiving a minimum of an a priori defined frequency of infusions for at least 45 weeks (85%) of the year under consideration"
4. Participant is willing and able to comply with the requirements of the protocol
5. Participant is proficient in the English language to allow for use of the Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) tool.

Exclusion Criteria:

1. Participants with an active Factor VIII (FVIII) inhibitory antibody (≥ 0.4 Bethesda units (BU) using the Nijmegen modification of the Bethesda assay or ≥ 0.6 BU using the Bethesda assay) at any time prior to screening
2. Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand's disease)
3. Participant has participated in a clinical study involving a medicinal product or device within 30 days prior to enrollment or is scheduled to participate in a clinical study involving a medical product or device during the course of this study
4. Participant is a family member or employee of the investigator

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with moderate to severe hemophilia A in the United States or Canada.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2016-11-02 (Actual); Study Completion 2016-11-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the response to the Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) outcomes tool | Baseline; weeks 6 and 12
  The GAS-Hem is an online instrument for setting and tracking personalized goals related to hemophilia. The GAS-Hem uses a 5-point scale to record the degree of attainment in relation to individually defined goal areas between an established baseline (scaled as -1) and follow-up time points (here, 6 weeks and 12 weeks). The scale range is +2 (much better outcome) to -2 (much worse outcome), where 0 represents the desired outcome. The process includes a facilitator to ensure that the outcome descriptions for the scale levels are reasonably attainable (not too hard or too easy) and represent roughly equivalent change between levels (ie scores). The overall scoring formula results in a summary score of 50 when all goals are attained (individual goal attainment = 0). Scores >50 indicate generally better than expected outcomes in goal attainment. Scores <50 indicate that, overall, goals were not achieved. The overall total scores range is dependent on the average number of goals.
Change from baseline of the measurement of the responsiveness (sensitivity to change) of GAS-Hem compared with the SF-36 | Baseline; weeks 6 and 12
  Comparison of outcomes on the Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) with the Medical Health Outcomes Study Health Survey Short Form-36 (SF-36) measures. The analysis will compare effect sizes calculated for the GAS-Hem and the SF-36 using Cohen's d and standardized response means.
Change from baseline of the measurement of the responsiveness (sensitivity to change) of GAS-Hem compared with the PedQL | Baseline; weeks 6 and 12
  Comparison of outcomes on the Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) with the Pediatric Quality of Life Inventory (PedsQL) measures. The analysis will compare effect sizes calculated for the GAS-Hem and the PedsQL using Cohen's d and standardized response means.

SECONDARY OUTCOMES:
Change from baseline of Quality of life (QoL) outcomes: Medical Health Outcomes Study Health Survey Short Form-36 (SF-36) | Baseline; weeks 6 and 12
  The SF-36 is a 36 item survey of physical functioning, role limitations (both physical and emotional), bodily pain, general health vitality, social functioning and mental health administered to adults aged 19 and older. The instrument measure health related quality of life on a scale of 0 (lowest level) to 100 (highest level).
Change from baseline of Quality of life (QoL) outcomes: Pediatric Quality of Life Inventory Version 4.0 Generic Core Scale (PedsQL) | Baseline; weeks 6 and 12
  The PedsQL is a 23 item survey that assesses physical functioning, emotional functioning, social functioning, and school functioning in children and adolescents aged 5 to 18. The PedsQL measures health related quality of life on a scale of 0 (lowest quality of life) to 100 (highest quality of life).
Participant perception of the GAS-Hem as a useful means of identifying and monitoring change in relevant goal areas | Week 12
  Measured using a questionnaire to test acceptability and usefulness of Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) to patients, and where applicable to their parents or guardians.
Clinician perception of the GAS-Hem as a useful means of monitoring clinical progress in patient identified goal areas | Week 12
  Measured using a questionnaire for clinicians designed to test their perception of the usefulness of Standardized Goal Attainment Scaling menu for Hemophilia (GAS-Hem) for monitoring clinical progress.
Number and Location of Bleeds | Within six months prior starting study through week 12 in the study
  History of bleeding episodes in the six months prior to signing informed consent will be collected. Participants will record details of each subsequent bleeding episode in the participant diary during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (4):
- United States (2):
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Oregon Health & Science University, Portland, Oregon
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc14db2bf003ab45660